CLINICAL TRIAL: NCT04377087
Title: Phase IIA Trial of Delayed Initiation of Olaparib Maintenance Therapy in Platinum Sensitive Recurrent Ovarian Cancer
Brief Title: Delayed Initiation of Olaparib Maintenance Therapy in Platinum Sensitive Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Sarah E Taylor (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor-Investigator, Sarah E Taylor, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 19-164
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer
Keywords: PARP-I; BRCA mutation; Epithelial ovarian cancer (EOC); Olaparib; platinum sensitive; recurrent ovarian carcinoma; Poly ADP-Ribose Polymerase (PARP) inhibitor.
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Olaparib (Experimental): Olaparib dosed at 300mg orally twice daily, started when CA125 rises by two-fold of nadir value.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib is a potent oral poly (ADP-ribose) polymerase (PARP) inhibitor that induces synthetic lethality in BRCA1/2 deficient tumor cells through the formation of double-stranded DNA breaks which cannot be accurately repaired, which leads to disruption of cellular homeostasis and cell death.
  Other Names: Lynparza™

SUMMARY:
The purpose of this study is to test if delaying the start of the olaparib until there is a rise in a tumor marker called CA-125 will result in a longer time until the next or different treatment for the patient's cancer. The study will also evaluate how delaying the start of maintenance therapy will affect symptoms; physical functioning; quality of life; and impact on finances.

DETAILED DESCRIPTION:
This is a Phase II trial will investigate if waiting until the time of chemical recurrence, denoted by rising CA125, to start a PARP inhibitor will lead to an improved time to next therapy with improved quality of life and at a lower financial toxicity.

PARP-I have shown efficacy as both monotherapy and as maintenance therapy. This trial will explore whether patients with recurrent ovarian cancer could derive the same efficacy benefit from a delayed start of a PARP-I compared to immediate maintenance therapy. Delayed start would have the benefit of sparing the physical, psychological, and financial toxicity associated with prolonged treatment. This approach would be particularly relevant in a population of platinum-sensitive patients who can have prolonged treatment-free intervals.

With widespread use of PARP-I, regardless of timing, understanding, and overcoming PARP-I resistance is becoming a major clinical need.

Enrollment will start within 8 weeks of completion of platinum-based treatment. Monitored with CA 125 levels every 28 days. Olaparib will be started when CA 125 rises by two-fold of their nadir value. Olaparib will be dosed at 300 mg orally twice a day, 28 days of treatment will be a cycle. Follow-up will consist of CA125 drawn every 28 days and CT scans obtained at doubling of CA- 125 and then every 12 weeks* to assess for recurrence or progression. Clinician- and patient-reported adverse events recorded every 28 days. Cancer-related worry and distress assessed every 28 days. Measures of quality of life and physical function, and financial toxicity assessed every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient has platinum-sensitive, recurrent ovarian, fallopian-tube or peritoneal cancer. Platinum sensitivity is defined as complete clinical remission after frontline chemotherapy lasting greater than 6 months
* Patient has completed at least 2 courses of platinum-based chemotherapy with a PR or CR as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.139 or a CA-125 response, according to Gynecological Cancer InterGroup (GCIG) criteria40
* BRCA testing required (results not needed for registration)
* ECOG performance status score of 0, 1, or 2 (See Appendix A)
* Life expectancy greater than 6 months
* Normal organ and marrow function as defined: Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelets ≥ 100 x 109/L; Hemoglobin (Hgb) ≥ 8 g/dL (blood transfusions to reach this amount are allowed); Serum creatinine ≤ 1.5 mg/dL; Total serum bilirubin ≤ 1.5 x ULN; AST and ALT ≤ 2.5 x ULN
* Able to take oral medication
* Not pregnant and not breastfeeding
* Able to understand and willingness to sign a written informed consent document
* Patients must be enrolled within 8 weeks of completing last cycle of chemotherapy

Exclusion Criteria:

* Patient has had a prior invasive malignancy diagnosed within the last five years (except [1] non-melanoma skin cancer or [2] prior in situ carcinoma of the cervix or breast [3] has been without evidence of invasive disease for greater than 3 years)
* Patients receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib
* Uncontrolled intercurrent illness that could affect their participation in the study including, but not limited to, ongoing or active infection; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; known inadequately controlled hypertension; significant pulmonary disease including dyspnea at rest, patients requiring supplemental oxygen, or poor pulmonary reserve; or psychiatric illness/social situations that would limit compliance with study requirements
* Impairment of gastrointestinal function or disease that may significantly alter the absorption of olaparib
* Patients who have received prior treatment with a PARP inhibitor
* History of noncompliance to medical regimens

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecological cancers
Enrollment: 3 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Taylor, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olaparib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Olaparib
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 63.7 [52 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Next Therapy
Description: The time to next therapy from completion of platinum-based therapy for treatment of recurrence until initiation of post-olaparib treatment.
Time Frame: Up to 35 months
Population: All enrolled participants that received a subsequent therapy.
Measure: Number; unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 2
months
  Patient 2: number analyzed (Participants) | 1
  Patient 2 | 1
  Patient 3: number analyzed (Participants) | 1
  Patient 3 | 3

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) defined as time from enrollment until detected recurrence or progression of disease, via Response Evaluation Criteria in Solid Tumors , or death from any cause.. Per RECIST 1.1, Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 35 months
Population: All enrolled participants that had radiologically confirmed disease progression.
Measure: Number; unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 1
months | 3

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival as defined as the time from enrollment to death from any cause.
Time Frame: Up to 35 months
Population: Participants that experienced the event of death.
Measure: Number; unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 1
months | 15

4. Secondary Outcome: Overall Response Rate (ORR)
Description: The proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 35 months
Population: Zero treated patients that experienced a radiologically measurable complete or partial response per RECIST v1.1
Arm/Group | Olaparib
Number analyzed (Participants) | 0

5. Secondary Outcome: The Functional Assessment of Cancer Therapy + Ovarian-specific Scale (FACT-O)
Description: Health-related quality of life measured via The Functional Assessment of Cancer Therapy + Ovarian-specific scale (FACT-O). The FACT-O includes a list of statements that [other] people with ovarian cancer have said are important. The patient is asked to circle or mark one number per line to indicate their response as it applies to the prior 7 days. The scoring ranges from 0 (Not at all) to 4 (very much).
Time Frame: Up to 37 months
Population: Longitudinal assessments unavailable per limited enrollment. No data collected.
Arm/Group | Olaparib
Number analyzed (Participants) | 0

6. Secondary Outcome: PROMIS Physical Function-20a
Description: Physical function assessed through the PROMIS Physical Function-20a assesses self-reported performance of physical activities. The PROMIS includes a list of statements related to physical performance, with scores of 0 (Always) to 5 (Rarely).
Time Frame: Up to 35 months
Population: Longitudinal assessments unavailable per limited enrollment. No data collected.
Arm/Group | Olaparib
Number analyzed (Participants) | 0

7. Secondary Outcome: Assessment of Survivor Concerns (ASC) Worry Subscale and Impact of Event Scale (IES-R)
Description: The Assessment of Survivor Concerns (ASC) Worry Subscale and Impact of Event Scale (IES-R) will be used to measure worry and distress. The assessment includes a list of statements related to worry and stress experience during the patients prior, with responses ranging from 0 (Not at all) to 4 (Extremely). This assessment includes three subscales, the Intrusion subscale, the Avoidance subscale and the Hyperarousal subscale, which are each related to specific questions.
Time Frame: Up to 35 months
Population: Longitudinal assessments unavailable per limited enrollment. No data collected.
Arm/Group | Olaparib
Number analyzed (Participants) | 0

8. Secondary Outcome: Modified Collection of Indirect and Non-medical Direct Costs (COIN)
Description: Financial toxicity measured through (a) monetary measure using the Modified Collection of Indirect and Non-medical Direct Costs (COIN), (b) objective measure of financial burden assessed using Barrera et al's Economic Hardship questionnaire, and (c) subjective measure of financial distress will be gauged using the Comprehensive Score for Financial Toxicity (COST Measure).
Time Frame: Up to 35 months
Population: Longitudinal assessments unavailable per limited enrollment. No data collected.
Arm/Group | Olaparib
Number analyzed (Participants) | 0

9. Secondary Outcome: Adverse Events Possibly, Probably or Definitely Related to Treatment
Description: The number of patients that experience Adverse Events per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 that were determined to be possibly, probably or definitely related to study treatment.
Time Frame: Up to 35 months
Population: Treated patients that experienced adverse events related to study treatment.
Measure: Number; unit: participants
Arm/Group | Olaparib
Number analyzed (Participants) | 2
participants
  Pruritus (non-serious) | 1
  Lymphocyte count decreased (non-serious) | 1
  Fatigue (non-serious) | 1

ADVERSE EVENTS:
Time Frame: Adverse Events collected for up to 35 months
Arm/Group | Olaparib
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib (N=3)
Hypertension (Vascular disorders) | 2
Renal calculi (Renal and urinary disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Fatigue (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT04377087/Prot_SAP_000.pdf